CLINICAL TRIAL: NCT06982404
Title: ZeroHeart Biopsy - Prediction of Deceased Donor Heart Transplant Performance From Organ Donors Using Pre-Transplant Biopsies - A Pilot Study
Acronym: ZeroHeart
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Alberta Transplant Applied Genomics Centre (Unknown)
Responsible Party: Principal Investigator, Roxana Moayedifar, MD PhD, Principal Investigator, Medical University of Vienna
Other Study IDs: 2032/2024
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Heart Transplantation; Graft Rejection; Myocardial Injury; Organ Preservation; Biopsy; Gene Expression Profiling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Right ventricular myocardial tissue biopsies will be obtained from donor hearts at the time of organ procurement ("Time Zero"). Each biopsy will be divided into two parts: one part will be processed for routine histopathology, and the other will be preserved in RNAlater® for molecular analysis, including gene expression profiling. These tissue samples may also be used for future DNA and RNA extraction and related analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Time Zero Donor Heart Biopsy for Molecular Analysis — This intervention involves obtaining a right ventricular myocardial biopsy from the donor heart at the time of organ procurement ("Time Zero"), prior to transplantation. The biopsy is divided into two parts: one for routine histopathological evaluation and the other preserved in RNAlater® for molecular analysis using microarray technology. This molecular profiling is designed to detect early tissue injury and gene expression patterns associated with graft viability and transplant outcomes. The intervention is performed only once per donor and does not alter the standard clinical care of the recipient.

SUMMARY:
The goal of this observational study is to evaluate whether molecular analysis of donor heart biopsies taken at the time of organ removal ("Time Zero") can help predict the future function and rejection risk of the transplanted heart in adult transplant recipients.

The main questions it aims to answer are:

* Can early molecular injury in the donor heart, caused by brain death or circulatory death, be detected at the time of organ removal?
* Can these early molecular findings predict short-, mid-, and long-term transplant outcomes, such as graft function or rejection?

Participants will:

* Include heart donors whose hearts are being transplanted (both standard and marginal donors, including DBD and DCD cases)
* Provide two small biopsies from the donor heart at the time of organ removal: one for routine pathology, one for microarray-based molecular analysis
* Have routine follow-up biopsies after transplantation as part of standard care (no additional procedures required beyond medical standard)

Researchers will compare biopsy results from different donor types (standard vs. marginal, DBD vs. DCD) to see if early molecular signals are linked to later heart transplant outcomes.

ELIGIBILITY:
Inclusion Criteria:

All hearts from standard and expanded criteria donors as well as donor hearts from Donation after circulatory death (DCD) undergoing a heart biopsy at pre-implantation (at procurement) will be included. Consent will be obtained from the recipient at the time of transplant listing.

Exclusion Criteria:

Hearts will be excluded from the study if the participating clinician decides to discard the organ before transplantation or the recipient declines that the biopsy will be performed at the organ procurement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in this study include deceased heart donors and their corresponding transplant recipients. Donors will include both standard criteria donors and expanded criteria donors, including donations after brain death (DBD) and donations after circulatory death (DCD). Right ventricular heart tissue biopsies will be obtained from these donors at the time of organ procurement. Follow-up data will be collected from the adult transplant recipients of these donor hearts, based on routine clinical care (e.g., biopsies, echocardiography, and medical records) over a 12-month post-transplant period.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of Post-Transplant Heart Function Based on Time Zero Molecular Biopsy Profiles | From enrollment to the end of follow-up at 12 months
  This outcome assesses whether gene expression patterns identified in right ventricular heart tissue biopsies taken at the time of organ procurement ("Time Zero") can predict the function of the transplanted heart over a 12-month period. The biopsies are analyzed using microarray technology to detect molecular signs of tissue injury or inflammation present before transplantation.
  Post-transplant heart function will be evaluated through:
  Routine endomyocardial biopsies performed at standard clinical timepoints (2 weeks, 1 month, 2 months, 3 months, 6 months, and 1 year) to assess for signs of graft rejection or injury
  Echocardiography to measure cardiac function (e.g., ejection fraction, wall motion)
  Clinical indicators such as the need for mechanical circulatory support or other interventions
  The goal is to determine whether specific molecular markers in the donor biopsy are associated with better or worse transplant outcomes, such as rejection episodes or reduced cardiac function

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Yes, anonymized individual participant data (IPD) collected during the study will be shared with qualified researchers upon reasonable request. The data will include molecular profiling results, clinical outcome measures, and associated metadata, and will be handled and stored by ATAGC (Alberta Transplant Applied Genomics Centre) in compliance with privacy regulations and ethical standards. All shared data will be fully de-identified to protect participant confidentiality. Requests for access will be reviewed and approved by the study's data access committee.
Supporting Information: Study Protocol, SAP, ICF, CSR